CLINICAL TRIAL: NCT06216821
Title: OPT-CAD Score Guided Dual Antiplatelet De-escalation Time in Patients With Acute Coronary Syndrome Undergoing Undergoing Percutaneous Coronary Intervention: a Register-based Randomized Controlled Study
Brief Title: OPT-CAD Score GUIded Dual ANtiplatelet De-esCalation Time
Acronym: OPT-GUIDNACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Yi Li, Professor, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPT-GUIDANCE V1.0
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard DAPT therapy (Active Comparator): Standard DAPT therapy for 12 mouths
  Interventions: Drug: standard DAPT
- OPT-CAD score guided de-escalation DAPT therapy (Experimental): Patients at moderate to high risk of ischemic events assessed by the OPT-CAD score will receive DAPT therapy for 3 months followed by P2Y12 inhibitor monotherapy for 9 months; Patients at low risk of ischemic events assessed by the OPT-CAD score will receive DAPT for 1 month follow by P2Y12 inhibitor monotherapy for 11 months.
  Interventions: Drug: OPT-CAD score guided DAPT de-escalation

INTERVENTIONS:
Drug: standard DAPT — standard DAPT with aspirin and a P2Y12 inhibitor for 12 months after DES implantation.
  Arms: Standard DAPT therapy
Drug: OPT-CAD score guided DAPT de-escalation — De-escalation DAPT at 3 months for moderate to high risk patients and de-escalation DAPT at 1 month for low risk patients.
  Arms: OPT-CAD score guided de-escalation DAPT therapy

SUMMARY:
Monotherapy with a P2Y12 inhibitor after a minimum period of DAPT following percutaneous coronary intervention (PCI) is an emerging de-escalation antiplatelet strategy in recent years. However, the optimal timing for de-escalating DAPT in ACS patients undergoing PCI remains debated. The OPT-CAD score is a risk stratification tool derived from Chinese patients which has been demonstrated superior predictive capabilities for ischemic events and all-cause mortality than the GRACE score. Therefore, we hypothesize that the OPT-CAD score can be used to guide the timing of the DAPT de-escalation strategy to monotherapy with P2Y12 inhibitors for ACS patients, that is, low-risk patients could be de-escalated after 1 month, while high-risk patients could be de-escalated after 3 months, so as to achieve individualized antithrombotic therapy and maximize patient benefit.

DETAILED DESCRIPTION:
Antiplatelet therapy is a cornerstone of secondary prevention in patients with coronary artery disease. However, as the use of more potent antithrombotic therapy, it not only lowers ischemic risk but increases bleeding. Therefore, fully balancing the risks of thrombosis and bleeding to maximize patient benefit is the basis for antiplatelet therapy. Although there are several scoring systems to assess the risk of thrombotic or bleeding, such as GRACE score, CRUSADE score, PARIS score, and ARC-HBR criteria, the value of the above scoring systems from western populations in guiding dual antiplatelet therapy (DAPT) decisions has not been confirmed. The previous guidelines recommend considering the PRECISE-DAPT score and DAPT score to guide DAPT duration, but their practical application remains limited. The 2020 ESC NSTE-ACS guidelines pointed out that there is still a gap between evidence and practice regarding whether risk-stratified treatment strategies can improve the prognosis of patients, which urgently requires randomized controlled trials (RCTs) for validation.

Monotherapy with a P2Y12 inhibitor after a minimum period of DAPT following percutaneous coronary intervention (PCI) is an emerging de-escalation strategy DAPT in recent years. Previous RCTs such as STOPDAPT-2, SMART-CHOICE, TICO, and TWILIGHT have demonstrated that compared with the conventional 12-month DAPT regimen, de-escalation of DAPT reduced the risk of bleeding without a significant increase in ischaemic events. To be specific, the intervention groups switched to ticagrelor monotherapy after 3 months of DAPT, resulting in comparable ischemic event rates among both TICO trial enrolled ACS patients undergoing PCI and TWILIGHT trial enrolled high-risk patients undergoing PCI. Meanwhile, when STOPDAPT-2 trial enrolled low-risk patients undergoing PCI, the results also indicated that clopidogrel monotherapy after 1 month of DAPT results in similar thrombotic event risks. However, when STOPDAPT-2 ACS trial enrolled ACS patients, compared to the 12-month DAPT group, the results showed that switching from 1- to 2-month DAPT to clopidogrel monotherapy resulted in an increased incidence of myocardial infarction. Given these findings, the optimal timing for de-escalation of DAPT in ACS patients undergoing PCI remain debated.

The Optimal antiPlatelet Therapy for Chinese patients with Coronary Artery Disease (OPT-CAD) score, a risk stratification tool derived from a real-world, multicenter registration study of Chinese patients, has better predictive performance for ischemic events and all-cause mortality at 1-year than those of The Global Acute Coronary Event Registration (GRACE) score. Through the analysis of OPT-CAD population, it was found that low-risk and medium-high risk patients with OPT-CAD scores accounted for about 2/3 and 1/3, respectively, and the risk of major adverse cardiovascular events (MACE) in medium-high risk patients at 1 year follow-up was about 3 times that of low-risk patients. Therefore, we hypothesize that the OPT-CAD score can be used to guide the timing of DAPT de-escalation strategy to monotherapy with P2Y12 inhibitors for ACS patients, that is, low-risk patients could be de-escalated after 1 month, while high-risk patients could be de-escalated after 3 months, so as to achieve individualized antithrombotic therapy and maximize patient benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with ages of 18-80 years;
2. Patients with clinically diagnosed ACS who have undergone at least one DES implantation;
3. Individuals capable of completing the OPT-CAD scoring calculation;
4. Researchers assessing that participants can tolerate at least a 12-month duration of DAPT therapy;
5. Written informed consent provided.

Exclusion Criteria:

1. Left main coronary artery lesion PCI;
2. Allergy to study drugs such as aspirin, clopidogrel, or ticagrelor;
3. Meeting 1 major or 2 minor criteria for high bleeding risk according to the ARC-HBR criteria;
4. Anticipated need for revascularization or surgical intervention within 12 months;
5. Severe ischemia or hemorrhage events during the current hospitalization;
6. Life expectancy of other serious diseases is less than 1 year;
7. Pregnant or women of childbearing age who intend to conceive within 1 year;
8. Participation in other clinical trials while still under observation;
9. Researchers considering ineligibility for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3490 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) | 12 months
  NACE is defined as a composite of all cause death, myocardial infarction, stroke, stent thrombosis or BARC type 2,3, 5 bleeding

SECONDARY OUTCOMES:
BARC type 2,3, or 5 bleeding | 3 months and 12 months
BARC type 3 or 5 bleeding | 3 months and 12 months
Major adverse cardiac and cerebral events (MACE) | 3 months and 12 months
  MACE is defined as a composite of all cause death, myocardial infarction, stent thrombosis or ischemic stroke
All cause death | 3 months and 12 months
Stent thrombosis | 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, PhD, Study Chair — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Kim BK, Hong SJ, Cho YH, Yun KH, Kim YH, Suh Y, Cho JY, Her AY, Cho S, Jeon DW, Yoo SY, Cho DK, Hong BK, Kwon H, Ahn CM, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y; TICO Investigators. Effect of Ticagrelor Monotherapy vs Ticagrelor With Aspirin on Major Bleeding and Cardiovascular Events in Patients With Acute Coronary Syndrome: The TICO Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2407-2416. doi: 10.1001/jama.2020.7580. PMID 32543684
- [Background] Mehran R, Baber U, Sharma SK, Cohen DJ, Angiolillo DJ, Briguori C, Cha JY, Collier T, Dangas G, Dudek D, Dzavik V, Escaned J, Gil R, Gurbel P, Hamm CW, Henry T, Huber K, Kastrati A, Kaul U, Kornowski R, Krucoff M, Kunadian V, Marx SO, Mehta SR, Moliterno D, Ohman EM, Oldroyd K, Sardella G, Sartori S, Shlofmitz R, Steg PG, Weisz G, Witzenbichler B, Han YL, Pocock S, Gibson CM. Ticagrelor with or without Aspirin in High-Risk Patients after PCI. N Engl J Med. 2019 Nov 21;381(21):2032-2042. doi: 10.1056/NEJMoa1908419. Epub 2019 Sep 26. PMID 31556978
- [Background] Hahn JY, Song YB, Oh JH, Chun WJ, Park YH, Jang WJ, Im ES, Jeong JO, Cho BR, Oh SK, Yun KH, Cho DK, Lee JY, Koh YY, Bae JW, Choi JW, Lee WS, Yoon HJ, Lee SU, Cho JH, Choi WG, Rha SW, Lee JM, Park TK, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC; SMART-CHOICE Investigators. Effect of P2Y12 Inhibitor Monotherapy vs Dual Antiplatelet Therapy on Cardiovascular Events in Patients Undergoing Percutaneous Coronary Intervention: The SMART-CHOICE Randomized Clinical Trial. JAMA. 2019 Jun 25;321(24):2428-2437. doi: 10.1001/jama.2019.8146. PMID 31237645
- [Background] Watanabe H, Domei T, Morimoto T, Natsuaki M, Shiomi H, Toyota T, Ohya M, Suwa S, Takagi K, Nanasato M, Hata Y, Yagi M, Suematsu N, Yokomatsu T, Takamisawa I, Doi M, Noda T, Okayama H, Seino Y, Tada T, Sakamoto H, Hibi K, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Hanaoka KI, Morino Y, Kozuma K, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 Investigators. Effect of 1-Month Dual Antiplatelet Therapy Followed by Clopidogrel vs 12-Month Dual Antiplatelet Therapy on Cardiovascular and Bleeding Events in Patients Receiving PCI: The STOPDAPT-2 Randomized Clinical Trial. JAMA. 2019 Jun 25;321(24):2414-2427. doi: 10.1001/jama.2019.8145. PMID 31237644
- [Background] Watanabe H, Morimoto T, Natsuaki M, Yamamoto K, Obayashi Y, Ogita M, Suwa S, Isawa T, Domei T, Yamaji K, Tatsushima S, Watanabe H, Ohya M, Tokuyama H, Tada T, Sakamoto H, Mori H, Suzuki H, Nishikura T, Wakabayashi K, Hibi K, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Morino Y, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 ACS Investigators. Comparison of Clopidogrel Monotherapy After 1 to 2 Months of Dual Antiplatelet Therapy With 12 Months of Dual Antiplatelet Therapy in Patients With Acute Coronary Syndrome: The STOPDAPT-2 ACS Randomized Clinical Trial. JAMA Cardiol. 2022 Apr 1;7(4):407-417. doi: 10.1001/jamacardio.2021.5244. PMID 35234821
- [Background] Han Y, Chen J, Qiu M, Li Y, Li J, Feng Y, Qiu J, Meng L, Sun Y, Tao G, Wu Z, Yang C, Guo J, Pu K, Chen S, Wang X. Predicting long-term ischemic events using routine clinical parameters in patients with coronary artery disease: The OPT-CAD risk score. Cardiovasc Ther. 2018 Oct;36(5):e12441. doi: 10.1111/1755-5922.12441. Epub 2018 Jun 28. PMID 29869835
- [Background] Li X, Qiu M, Na K, Li Y, Ma S, Qi Z, Li J, Li Y, Han Y. Comparison of the efficacy and safety of ticagrelor and clopidogrel in patients with acute coronary syndrome after risk stratification. Catheter Cardiovasc Interv. 2021 May 1;97 Suppl 2:1032-1039. doi: 10.1002/ccd.29591. Epub 2021 Mar 2. PMID 33650763
- [Background] Zhao Y, Li J, Ma S, Jiang Z, Li Z, Wang X, Han Y, Li Y. Impact of extended dual antiplatelet therapy on long-term prognosis in patients with acute coronary syndrome complicated with anemia: A sub-analysis of the real-world OPT-CAD study. Catheter Cardiovasc Interv. 2021 Aug 1;98(2):E235-E242. doi: 10.1002/ccd.29676. Epub 2021 Apr 5. PMID 33817946
- [Background] Ma S, Jiang Z, Qiu M, Li Z, Bian L, Li Y, Han Y. Dual Antiplatelet Therapy Duration in Medically Managed Acute Coronary Syndrome Patients: Sub-Analysis of the OPT-CAD Study. Adv Ther. 2020 Jul;37(7):3150-3161. doi: 10.1007/s12325-020-01376-0. Epub 2020 May 16. PMID 32418142
- [Background] Wang H, Qi J, Li Y, Tang Y, Li C, Li J, Han Y. Pharmacodynamics and pharmacokinetics of ticagrelor vs. clopidogrel in patients with acute coronary syndromes and chronic kidney disease. Br J Clin Pharmacol. 2018 Jan;84(1):88-96. doi: 10.1111/bcp.13436. Epub 2017 Nov 3. PMID 28921624
- [Background] Han Y, Liao Z, Li Y, Zhao X, Ma S, Bao D, Qiu M, Deng J, Wang J, Qu P, Jiang C, Jia S, Yang S, Ru L, Feng J, Gao W, Huang Y, Tao L, Han Y, Yang K, Wang X, Zhang W, Wang B, Li Y, Yang Y, Li J, Sheng J, Ma Y, Cui M, Ma S, Wang X, Li Z, Stone GW. Magnetically Controlled Capsule Endoscopy for Assessment of Antiplatelet Therapy-Induced Gastrointestinal Injury. J Am Coll Cardiol. 2022 Jan 18;79(2):116-128. doi: 10.1016/j.jacc.2021.10.028. Epub 2021 Nov 6. PMID 34752902
- [Background] Li Y, Wang X, Bao D, Liao Z, Li J, Han X, Wang H, Xu K, Li Z, Stone GW, Han Y. Optimal antiplatelet therapy for prevention of gastrointestinal injury evaluated by ANKON magnetically controlled capsule endoscopy: Rationale and design of the OPT-PEACE trial. Am Heart J. 2020 Oct;228:8-16. doi: 10.1016/j.ahj.2020.06.004. Epub 2020 Jun 15. PMID 32745734
- [Background] Li Y, Jing Q, Wang B, Wang X, Li J, Qiao S, Chen S, Angiolillo DJ, Han Y. Extended antiplatelet therapy with clopidogrel alone versus clopidogrel plus aspirin after completion of 9- to 12-month dual antiplatelet therapy for acute coronary syndrome patients with both high bleeding and ischemic risk. Rationale and design of the OPT-BIRISK double-blinded, placebo-controlled randomized trial. Am Heart J. 2020 Oct;228:1-7. doi: 10.1016/j.ahj.2020.07.005. Epub 2020 Jul 9. PMID 32739652
- [Background] Han Y, Claessen BE, Chen SL, Chunguang Q, Zhou Y, Xu Y, Hailong L, Chen J, Qiang W, Zhang R, Luo S, Li Y, Zhu J, Zhao X, Cheng X, Wang J, Su X, Tao J, Sun Y, Wang G, Li Y, Bian L, Goel R, Sartori S, Zhang Z, Angiolillo DJ, Cohen DJ, Gibson CM, Kastrati A, Krucoff M, Mehta SR, Ohman EM, Steg PG, Liu Y, Dangas G, Sharma S, Baber U, Mehran R. Ticagrelor With or Without Aspirin in Chinese Patients Undergoing Percutaneous Coronary Intervention: A TWILIGHT China Substudy. Circ Cardiovasc Interv. 2022 Apr;15(4):e009495. doi: 10.1161/CIRCINTERVENTIONS.120.009495. Epub 2022 Mar 23. PMID 35317615